CLINICAL TRIAL: NCT02799485
Title: A Phase II Study of sEphB4-HSA in Kaposi Sarcoma
Brief Title: sEphB4-HSA in Treating Patients With Kaposi Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Vasgene Therapeutics, Inc (Industry); The Emmes Company, LLC (Industry); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-096; NCI-2015-00052 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 096 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC 096 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U01CA121947 (NIH)
Record Dates: First submitted 2016-02-09; First posted 2016-06-15 (Estimated); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Skin Kaposi Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (recombinant EphB4-HSA fusion protein) (Experimental): Patients receive recombinant EphB4-HSA fusion protein IV over 1 hour on days 1 and 15. Patients with disease progression after 2 or more courses who have not experienced toxicity may receive recombinant EphB4-HSA fusion protein IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of further disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Behavioral: Quality-of-Life Assessment; Biological: Recombinant EphB4-HSA Fusion Protein

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Behavioral: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Recombinant EphB4-HSA Fusion Protein — Given IV
  Other Names: sEphB4-HSA

SUMMARY:
This phase II trial studies recombinant EphB4-HSA fusion protein (EphB4-HSA) in treating patients with Kaposi sarcoma. Recombinant EphB4-HSA fusion protein may block the growth of blood vessels that provide blood to the cancer, and may also prevent cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the clinical response and toxicity of recombinant EphB4-HSA fusion protein (sEphB4-HSA) (at initial dosing of 15 mg/kg every 2 weeks) in participants with Kaposi sarcoma.

SECONDARY OBJECTIVES:

I. To assess the safety of sEphB4-HSA in participants with Kaposi sarcoma (KS). II. To determine trough level exposure of sEphB4-HSA and correlate with tumor response.

III. To characterize the pharmacodynamics of sEphB4-HSA and correlate these effects with clinical response.

IV. Effects on viral replication and gene expression of human herpes virus-8 (HHV-8).

V. Changes in vascular endothelial growth factor (VEGF)-Notch-EphrinB2 angiogenic pathway.

VI. Effects on immune response and modulation. VII. Effects on tumor cell apoptosis and proliferation. VIII. Effects on sEphB4-HSA on human immunodeficiency virus (HIV) plasma viral loads in participants with HIV.

IX. To archive peripheral blood mononuclear cells (PBMCs) and tissue samples to be used in conjunction with samples collected in subsequent trials of sEphB4-HSA for future studies including identification of biomarkers predictive of response.

X. To evaluate the clinical response and toxicity of sEphB4-HSA (at increased dosing of 10 mg/kg every week) in participants with KS.

TERTIARY OBJECTIVES:

I. Describe baseline quality of life (QOL) scores, using the functional assessment of HIV Infection (FAHI) + Kaposi sarcoma (KS) questionnaire, in participants with KS, and explore changes in QOL of participants on treatment with sEphB4-HSA.

OUTLINE:

Patients receive recombinant EphB4-HSA fusion protein intravenously (IV) over 1 hour on days 1 and 15. Patients with disease progression after 2 or more courses who have not experienced toxicity may receive recombinant EphB4-HSA fusion protein IV over 1 hour on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of further disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 month; patients with partial response or better are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants may be treatment naïve, refractory to or intolerant of one or more prior therapies, or treated with prior systemic treatment including but not limited to liposomal doxorubicin
* Participants must have biopsy-proven KS involving skin with or without visceral involvement
* If HIV-positive, any cluster of differentiation (CD)4 count will be allowed on study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 or Karnofsky performance score (KPS) >= 60%
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 1,500/mcL*

  * Participants may be receiving growth factor support to meet these criteria
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Creatinine within normal institutional limit for the reference lab OR creatinine clearance >= 60 mL/min/1.73 m^2 as calculated by Cockcroft-Gault formula for participants with creatinine levels above institutional normal
* Participants must have cutaneous lesion(s) amenable to four (4) 5-mm tumor biopsies during the study (either 4 separate lesions measuring >= 5 mm each OR 2 separate lesions measuring >= 10 mm each) and at least five additional lesions measurable for assessment with no improvement over the past month
* Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 14 days prior to enrollment and again within 24 hours prior to starting cycle 1 of sEphB4-HSA; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME during receipt of sEphB4-HSA, and 12 weeks after discontinuation of sEphB4-HSA; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Documentation of HIV status; if participant is HIV positive, HIV-1 infection, as documented by any federally approved, licensed HIV rapid test performed in conjunction with screening (or enzyme-linked immunosorbent assay [ELISA], test kit, and confirmed by Western blot or other approved test); alternatively, this documentation may include a record demonstrating that another physician has documented the participant's HIV status based on either: 1) approved diagnostic tests, or 2) the referring physician's written record that HIV infection was documented, with supporting information on the participant's relevant medical history and/or current management of HIV infection

  * If the participant is HIV negative, documentation of a negative result for any federally approved, licensed HIV rapid test within 4 weeks prior to study enrollment will suffice; if the initial rapid test is positive, further approved confirmatory test results must be present to document the subject's HIV status
* If participant is HIV positive, participants must be on a stable antiretroviral regimen for at least 12 weeks prior to study enrollment
* There should be no evidence for improvement in KS in the 3 months prior to study enrollment, unless there is evidence for progression of KS in the 4 weeks immediately prior to study enrollment
* Participants must, in the opinion of the investigator, be capable of complying with the protocol

Exclusion Criteria:

* Inability to understand and inability to provide informed consent
* Participants who are receiving any other investigational agents
* Participants who have had anti-neoplastic treatment for KS (including chemotherapy, radiotherapy, local treatment including topical fluorouracil [5-FU], biological therapy or investigational therapy) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study OR those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Participants with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sEphB4-HSA or other agents used in study
* Participants who refuse antiretroviral therapy for HIV, if HIV positive
* Concurrent, acute, active infection, or treatment for infection, other than oral thrush or genital herpes, within 14 days of enrollment
* Participants for whom front-line cytotoxic therapy is indicated (i.e. symptomatic visceral or pulmonary KS or symptomatic KS impairing functional status)
* Concurrent neoplasia requiring cytotoxic therapy
* Participant is =< 2 years free of another primary malignancy; exceptions include the following:

  * Basal cell skin cancer
  * Cervical carcinoma in situ
  * Anal carcinoma in situ
* Any steroid treatment except for that required for replacement therapy in adrenal insufficiency, topical or injected testosterone for hypogonadism, or inhaled steroids for the treatment of asthma
* Previous local therapy of any KS-indicator lesion unless the lesion has clearly progressed since that local treatment; any prior local treatment to indicator lesions regardless of the elapsed time should not be allowed unless there is evidence of clear-cut progression of said lesion
* Female participants who are pregnant, lactating, or breast-feeding
* Breastfeeding should be discontinued if the mother is treated with sEphB4-HSA
* Participants with a recent history (< 6 months) of a major infarct including but not inclusive to bowel ischemia, cerebral vascular accident, transient ischemic attack, myocardial infarction, limb ischemia, or skin necrosis
* Participants with a QTcF (Fridericia correction formula) > 480 ms on 2 out of 3 electrocardiograms (EKGs) (if first EKG is < 480, no need to repeat, if first EKG is > 480 repeat twice for a total of 3 EKGs)
* Participants with uncontrolled sustained hypertension which will be defined as systolic blood pressure > 140, and diastolic blood pressure > 90, even with use of anti-hypertensive medications
* Participants with a recent history (< 6 months) of a major bleed which will be defined as a symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a fall in hemoglobin level 2 grams/dL or more, or leading to transfusion of two or more units of whole blood or packed red cells
* Participants on any dose of warfarin or are on full dose anticoagulation with other agents including low molecular weight heparin, antithrombin agents, antiplatelet agents and full dose aspirin within 7 days prior to study enrollment; participants on prophylactic doses of low molecular weight heparin and low dose anticoagulants are allowed.
* Cardiac related illnesses including, but not limited to:

  * Symptomatic congestive heart failure including participants with grade III/IV cardiac disease as defined by the New York Heart Association functional criteria
  * Unstable angina pectoris
  * Cardiac arrhythmia
* Proteinuria as defined as > 2+ on urine dipstick; if dipstick urinalysis shows >= 2+ proteinuria, 24-hour urine for protein must be < 2 grams
* Participants with diabetes mellitus with ketoacidosis or chronic obstructive pulmonary disease (COPD) requiring hospitalization in the preceding 6 months, or any other intercurrent medical condition that contraindicates treatment with sEphB4-HSA or places the participant at undue risk for treatment related complications
* Physical or psychiatric illness/social situations that in the estimation of the investigator would limit compliance with study requirements or place the participant at high risk of toxicity or non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Proportion of participants experiencing clinical response | 4 weeks (after 2 courses) and up to 12 months (end of follow-up)
  The observed proportions of participants experiencing clinical response and unacceptable toxicity will be calculated with 95% confidence intervals. For clinical response, the Kaplan-Meier method will be used to estimate the distribution for time to death assessed for up to 1 month after treatment completion; for time to progression assessed from chemotherapy initiation to first documented progression up to 1 month after treatment completion; and for time to response assessed from the first dose until first documented response up to 1 month after completion of treatment. The Kaplan-Meier method will then be used to estimate the distribution of time to response, time to relapse, and time to death. Time to response is the time from the first dose until documented first response. Time to progression is the time from first dose to first documented progression. Response duration is the time from first documented response to first documented progression.
Proportion of participants experiencing unacceptable toxicity | Up to 12 months (end of follow-up)
  Adverse events will be tabulated according to type and severity.

SECONDARY OUTCOMES:
Pharmacodynamic parameters of recombinant EphB4-HSA fusion protein | Days 1 and 15 of courses 1 and 2; days 1, 8, 15, and 22 of 1st 2 courses at escalated dose
  Descriptive statistics and graphical displays will be used to evaluate correlation between response and pharmacodynamics of EphB4-HSA. Depending on the number enrolled, the association between clinical response and changes in trough levels, pharmacodynamic endpoints, viral copy number, protein expression and activation status, and finally immune cell counts and activation status will be investigated using the nonparametric Wilcoxon rank sum test.
Trough levels of recombinant EphB4-HSA fusion protein | Days 1 and 15 of courses 1 and 2; days 1, 8, 15, and 22 of 1st 2 courses at escalated dose
  Descriptive statistics and graphical displays will be used to evaluate correlation between response and trough levels of EphB4-HSA. Depending on the number enrolled, the association between clinical response and changes in trough levels, pharmacodynamic endpoints, viral copy number, protein expression and activation status, and finally immune cell counts and activation status will be investigated using the nonparametric Wilcoxon rank sum test.

OTHER OUTCOMES:
Overall quality of life, assessed using the KS Functional Assessment of HIV questionnaire | Baseline, day 1, day 1 of course 4, 12 months (end of study)
  Five measures of overall quality of life will be scored: physical well-being, emotional well-being, functional and global well-being, social well-being, and cognitive functioning. For KS-specific symptoms, responses may be dichotomized to reflect positive or negative impact of these symptoms. General estimating equations using a log-binomial model will be used to assess changes in these symptoms over time.

CONTACTS AND LOCATIONS:
Overall Officials: Ida Wong-Sefidan, Principal Investigator — AIDS Malignancy Consortium
Locations (9):
- United States (9):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCSD Moores Cancer Center, La Jolla, California
  - UCLA CARE Center, Los Angeles, California
  - University of Miami, Miami, Florida
  - Grady Health System, Atlanta, Georgia
  - John H. Stroger Jr., Hospital of Cook County, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No